CLINICAL TRIAL: NCT07128901
Title: A Comparative Analysis of Lower-Limb Exoskeleton Technology for Non-Ambulatory Individuals With Spinal Cord Injury
Brief Title: Lower-Limb Exoskeleton Technology for Non-Ambulatory Individuals With Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: Shepherd Center, Atlanta GA (Other)
Responsible Party: Principal Investigator, Maegan Tucker, Assistant Professor, Georgia Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2331046-1
Record Dates: First submitted 2025-08-06; First posted 2025-08-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injuries
Keywords: lower limb exoskeleton
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Self-balancing lower limb exoskeleton (Experimental): Participants will use the self-balancing lower limb exoskeleton for 5 walking sessions and then complete a test session.
  Interventions: Device: Wandercraft Atalante X
- User-balancing lower limb exoskeleton (Experimental): Participants will use the user-balancing lower limb exoskeleton for 5 walking sessions and then complete a test session.
  Interventions: Device: Ekso Indego Therapy

INTERVENTIONS:
Device: Ekso Indego Therapy — User-balancing lower Limb exoskeleton
  Arms: User-balancing lower limb exoskeleton
Device: Wandercraft Atalante X — Self-balancing lower limb exoskeleton
  Arms: Self-balancing lower limb exoskeleton

SUMMARY:
The purpose of this study is to compare two types of wearable lower-extremity exoskeletons -a self-balancing device lower-extremity exoskeleton and a user-balancing device lower-extremity exoskeleton-to better understand their effects on the physiological responses to walking and the user experience in people with spinal cord injury.

DETAILED DESCRIPTION:
Although Lower Limb Exoskeleton technology holds promise for improving mobility and independence in people with Spinal Cord Injury, limited research has examined the physiological and psychological effects of walking with self-balancing lower limb exoskeleton technology compared to systems that require user-operated assistive aids. Moreover, no studies to date have directly compared the short- and long-term outcomes of two lower limb exoskeleton technology types: (1) self-balancing and (2) user-balancing. To address this gap, this study will conduct a head-to-head comparison of self-balancing and user-balancing lower limb exoskeleton technology in individuals with motor-complete (ASIA Impairment Scale Classification [AIS] A/B) Spinal Cord Injury-a population that remains underrepresented in rehabilitation robotics research despite advances in the field.

Study participants will complete 5 walking sessions and 2 test sessions with two different exoskeleton devices in a randomized order. During each test session, data will be collected using motion sensors, portable metabolic monitors, and muscle sensors.

ELIGIBILITY:
Inclusion Criteria:

* Subacute to chronic SCI (≥ 3mths post injury)
* Motor-complete (ASIA Impairment Scale classification A/B)
* Injury level T3-T11
* Age 18-70 yrs
* Height between 5'1" and 6'1"
* Weight <200 lbs (90kg)
* Seated hip width < 42cm
* Standing tolerance > 15mins
* Have sufficient upper limb strength to use a platform rolling walker, rolling walker, or forearm crutches
* Currently medically cleared and enrolled in the Shepherd Center Beyond Therapy program
* Medically cleared for weight-bearing activities
* Able to follow directions to safely participate in assessments

Exclusion Criteria:

* Existing skin lesions or wounds
* Hip or knee contracture > 10 degrees or ankle contracture > 5 degrees
* Severe or uncontrolled spasticity
* Non-healing fractures
* Uncontrolled autonomic dysreflexia
* Heart or peripheral vascular condition
* Pregnancy
* Active heterotopic ossification
* Active deep vein thrombosis
* Cognitive deficits that make it difficult for participants to follow verbal instructions or making it unsafe to participate in assessments.
* Any reason the principal investigator feels the potential participant may not be safe to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
10 meter walk test (10MWT) | 1 year
  This will be measured as the participant walks a distance of 10 meters at their self-selected (or comfortable) walking speed. Three 10-meter walk trials will be completed by each participant at each time point. The average of three 10MWT walking speeds will be analyzed and reported. This measure will be recorded in seconds and converted to meters/s with higher values indicating faster speed and lower values indicating slower speeds. Self-selected walking speed is highly correlated with functional ability and dependence.
6 minute walk test (6MWT) | 1 year
  This is a measurement of endurance and functional ability that assesses the participants ability to walk a distance (meters) over a time period of 6 minutes. It is measured in distance with greater distances indicating improved levels of endurance and functional ability.

SECONDARY OUTCOMES:
Neuromuscular activation of specified muscles | 1 year
  Electromyography sensors will measure the magnitude of muscle activation for the torso throughout the gait cycle. The average magnitude will be computed by averaging the time-series data across gait cycles and computing the average magnitude for the average gait cycle.
Walking economy | 1 year
  Walking economy is a measure of the energy cost of walking, quantified as the amount of oxygen consumed per kilogram of body weight per meter walked. It reflects the metabolic efficiency of gait, with lower values indicating more efficient walking. This measure will be obtained using the Cosmed K5 indirect calorimetry system during steady-state walking.
Rating of Perceived Exertion | 1 year
  The Rating of Perceived Exertion is a subjective measure of exertion based on an individual's perception of effort and fatigue during physical activity. The scale ranges from 6 (no exertion) to 20 (maximal exertion).
Total hemoglobin concentration | 1 year
  Total hemoglobin concentration refers to the amount of hemoglobin present in a given volume of blood. It is an indicator of muscle oxygenation dynamics. This measure will be obtained using continuous wave near-infrared spectroscopy.
User-experience survey | 1 year
  A custom survey will be administered to assess participant opinion on exoskeleton comfort, ease of use, perceived effort and overall satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- The Shepherd Center, Atlanta, Georgia, United States